CLINICAL TRIAL: NCT04954586
Title: Feasibility of Pain Informed Movement for People With Knee Osteoarthritis
Brief Title: Feasibility of Pain Informed Movement for Knee OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: The Arthritis Society, Canada (Other)
Responsible Party: Principal Investigator, Lisa Carlesso, Dr., McMaster University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pain Informed Movement
Record Dates: First submitted 2021-06-18; First posted 2021-07-08 (Actual); Results first posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-07

CONDITIONS: Knee Osteoarthritis
Keywords: Pain Management; Pain Modulation; Yoga; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pain Informed Movement (Experimental): This will be an 8-week in-person group exercise program held twice weekly, in which participants will receive pain Informed movement (60 minutes), with instructions provided for a third home session. Home sessions will be facilitated by exercise handout sheets. Pain education will be delivered through weekly access to videos. The pain informed movement component has been developed by a team member and will be delivered by an experienced yoga teacher.
  Interventions: Other: Pain Informed Movement

INTERVENTIONS:
Other: Pain Informed Movement — Participants will attend a twice weekly exercise program.

SUMMARY:
The pain experience and its associated mechanisms in people with knee osteoarthritis (OA) are known to be complex and multidimensional. The current understanding of OA pain mechanisms is incomplete, resulting in limited pain management strategies. There is high-quality evidence that suggests the use of exercise for people with knee OA can provide a reduction in pain, changes in quality of life, and have modest improvements in physical function. There is promising evidence to support that yoga for those with knee OA may improve pain intensity, function, and stiffness. The aim of this study is to establish the feasibility of a pain informed movement program, in addition to education for improving pain modulation. The data collected will be used to inform a pilot and feasibility randomized controlled trial (RCT) prior to a multi site RCT to assess the program's effectiveness with the primary outcome of change in pain severity mediated by change in descending modulation.

DETAILED DESCRIPTION:
Background

Exercise is regularly utilized as a first-line treatment for knee osteoarthritis, and its use is supported by high quality evidence to improve pain and function. Reductions in perceived pain can be explained in part by exercised-induced analgesia, which is thought to be mediated via numerous endogenous pathways. Furthermore, decreased nervous system sensitivity to noxious stimuli seem to play a role in the decreased pain experience of individuals who engage in exercise. These mechanisms likely play a role in improved function and reduced pain along with the improved balance, muscle strength and flexibility that are conventionally associated with exercise. In recent years multiple guidelines for non-surgical management of knee OA have begun to include mind-body therapies, such as yoga or tai-chi, as conditional or core treatment recommendations. Structured yoga programs have been shown to result in decreased pain and improved function when compared to no exercise and conventional exercise.

BDNF is a neurotrophin that appears to play an important role in the central modulation of pain in adults, and altered expression of BDNF is likely to play an important role in the pathophysiology of chronic pain. Individuals with knee OA have been shown to possess altered levels of serum BDNF compared to healthy controls, indicating that BDNF may be implicated in the pain-experience of patients with knee OA. Thus, BDNF has been identified as a therapeutic target in the treatment of pain resulting from central sensitization.

NGF is a neurotrophin known to play a critical role in the proper development of the nervous system. Evidence indicates that NGF is also involved in the increased pain experience of many individuals via peripheral sensitization of nociceptive neurons. Therefore, NGF levels have been shown to be elevated in a wide variety of chronic pain conditions including knee OA. Anti-NGF therapies are being highly studied as they have significant potential to decrease pain and improve function in individuals with OA that do not respond to conventional analgesics.

Objectives

The aim of this study is to establish the feasibility of a pain informed movement program, in addition to education for improving pain modulation. The data collected will be used to inform a pilot and feasibility randomized controlled trial (RCT) prior to a multi site RCT to assess the program's effectiveness with the primary outcome of descending modulation as a mediator of change in pain severity.

Research questions

1. Is the pain informed movement and education program feasible in terms of recruitment rate, treatment adherence, timelines, data collection procedures, patient follow-up and resources required?
2. Is the pain informed movement and education program feasible in terms of patient's satisfaction and acceptability?

Study Population

A convenience sample of 15 adults will be sought and is adequate to evaluate the feasibility of the program.

Recruitment

Participants will be recruited through the email lists of the McMaster Physical Activity Centre of Excellence (PACE) community. Recruitment posters will also be included in the McMaster Institute for Research on Aging (MIRA) newsletter. In addition, we will place postings on both PACE and MIRA social media pages.

Setting

The in-person 8-week exercise program will be held twice weekly at McMaster University's Physical Activity Centre of Excellence (PACE) located in the Ivor-Wynne Centre. Participants will complete the pain assessment, and have blood drawn at PACE by PACE staff who are certified phlebotomists.

Assessment

As part of participation in the study, participants will be asked to attend an assessment at the beginning of the study, and once again upon completing the 8-week exercise program. Participants will undergo pain modulation (CPM) testing, and the 30 Second Sit to Stand Test to determine leg strength and endurance. Lastly, participants will have their blood drawn at the beginning and end of the study. Participants will then be asked to complete a series of questionnaires about their pain and mood.

Exit Survey and Focus Group

A satisfaction survey will be conducted at the end of the program to evaluate the a priori feasibility criteria. Participants who indicated upon initially consenting to the study that they would like to participate in a focus group, will be contacted. Qualitative data collection will be used to explore participants experience and perceptions of the feasibility and acceptability of the program. A focus group will be conducted using audio or video recording (using Zoom), lasting between 45-60 minutes.

Statistical Analysis Plan (SAP)

All quantitative analyses will be conducted using SPSS 26. Descriptive statistics will be used to report feasibility outcomes, and survey responses will be summarized (using descriptive statistics) to identify trends in patient-reported outcomes. Qualitative interviews will be analyzed using Thematic content analysis to identify suggestions for program modification. Line-by-line reading of the transcripts will be performed by the authors and thematic patterns will be explored. Once themes and patterns are identified, each meaningful segment of text will be assigned a conceptual code. When conceptual codes become saturated, authors will build pattern codes where specific dimensions of clinicians' experiences will be clustered into recurring themes. Once the codes and themes are developed, participant and clinician partners will be invited to contribute to blinded data analysis to broaden interpretations and provide feedback on the quotes and emergent themes.

ELIGIBILITY:
Inclusion Criteria:

* 40 years of age and over
* Have a diagnosis of knee OA by a physician
* or fulfill the NICE criteria for knee OA diagnosis
* Have an average pain intensity of ≥3/10 on a numeric pain scale

Exclusion Criteria:

* Cannot communicate in English
* Have inflammatory arthritis or other systemic conditions
* Have had lower limb trauma
* Had surgery within the past 6-month, have participated in a similar knee OA exercise program in the prior 3-months
* Have used oral corticosteroids or had a corticosteroid injection in the index knee within 6-months prior to baseline assessment.
* Does not have access to the internet

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2022-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Carlesso, PhD, Principal Investigator — McMaster University
Locations (1):
- PACE, McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Fransen M, McConnell S, Harmer AR, Van der Esch M, Simic M, Bennell KL. Exercise for osteoarthritis of the knee: a Cochrane systematic review. Br J Sports Med. 2015 Dec;49(24):1554-7. doi: 10.1136/bjsports-2015-095424. Epub 2015 Sep 24. PMID 26405113
- [Background] Bannuru RR, Osani MC, Vaysbrot EE, Arden NK, Bennell K, Bierma-Zeinstra SMA, Kraus VB, Lohmander LS, Abbott JH, Bhandari M, Blanco FJ, Espinosa R, Haugen IK, Lin J, Mandl LA, Moilanen E, Nakamura N, Snyder-Mackler L, Trojian T, Underwood M, McAlindon TE. OARSI guidelines for the non-surgical management of knee, hip, and polyarticular osteoarthritis. Osteoarthritis Cartilage. 2019 Nov;27(11):1578-1589. doi: 10.1016/j.joca.2019.06.011. Epub 2019 Jul 3. PMID 31278997
- [Background] Cheung C, Wyman JF, Bronas U, McCarthy T, Rudser K, Mathiason MA. Managing knee osteoarthritis with yoga or aerobic/strengthening exercise programs in older adults: a pilot randomized controlled trial. Rheumatol Int. 2017 Mar;37(3):389-398. doi: 10.1007/s00296-016-3620-2. Epub 2016 Dec 2. PMID 27913870
- [Background] Simao AP, Mendonca VA, de Oliveira Almeida TM, Santos SA, Gomes WF, Coimbra CC, Lacerda AC. Involvement of BDNF in knee osteoarthritis: the relationship with inflammation and clinical parameters. Rheumatol Int. 2014 Aug;34(8):1153-7. doi: 10.1007/s00296-013-2943-5. Epub 2014 Jan 9. PMID 24399456
- [Background] Stoppiello LA, Mapp PI, Wilson D, Hill R, Scammell BE, Walsh DA. Structural associations of symptomatic knee osteoarthritis. Arthritis Rheumatol. 2014 Nov;66(11):3018-27. doi: 10.1002/art.38778. PMID 25049144
- [Background] Nijs J, Meeus M, Versijpt J, Moens M, Bos I, Knaepen K, Meeusen R. Brain-derived neurotrophic factor as a driving force behind neuroplasticity in neuropathic and central sensitization pain: a new therapeutic target? Expert Opin Ther Targets. 2015 Apr;19(4):565-76. doi: 10.1517/14728222.2014.994506. Epub 2014 Dec 18. PMID 25519921
- [Background] Kolasinski SL, Neogi T, Hochberg MC, Oatis C, Guyatt G, Block J, Callahan L, Copenhaver C, Dodge C, Felson D, Gellar K, Harvey WF, Hawker G, Herzig E, Kwoh CK, Nelson AE, Samuels J, Scanzello C, White D, Wise B, Altman RD, DiRenzo D, Fontanarosa J, Giradi G, Ishimori M, Misra D, Shah AA, Shmagel AK, Thoma LM, Turgunbaev M, Turner AS, Reston J. 2019 American College of Rheumatology/Arthritis Foundation Guideline for the Management of Osteoarthritis of the Hand, Hip, and Knee. Arthritis Rheumatol. 2020 Feb;72(2):220-233. doi: 10.1002/art.41142. Epub 2020 Jan 6. PMID 31908163
- [Background] Da Silva Santos R, Galdino G. Endogenous systems involved in exercise-induced analgesia. J Physiol Pharmacol. 2018 Feb;69(1):3-13. doi: 10.26402/jpp.2018.1.01. Epub 2018 May 8. PMID 29769416
- [Background] Galdino G, Romero T, Pinho da Silva JF, Aguiar D, de Paula AM, Cruz J, Parrella C, Piscitelli F, Duarte I, Di Marzo V, Perez A. Acute resistance exercise induces antinociception by activation of the endocannabinoid system in rats. Anesth Analg. 2014 Sep;119(3):702-715. doi: 10.1213/ANE.0000000000000340. PMID 24977916
- [Background] Koltyn KF, Arbogast RW. Perception of pain after resistance exercise. Br J Sports Med. 1998 Mar;32(1):20-4. doi: 10.1136/bjsm.32.1.20. PMID 9562159
- [Background] Esser S, Bailey A. Effects of exercise and physical activity on knee osteoarthritis. Curr Pain Headache Rep. 2011 Dec;15(6):423-30. doi: 10.1007/s11916-011-0225-z. PMID 21956792
- [Background] Ghasemi GA, Golkar A, Marandi SM. Effects of hata yoga on knee osteoarthritis. Int J Prev Med. 2013 Apr;4(Suppl 1):S133-8. PMID 23717763
- [Background] Merighi A, Salio C, Ghirri A, Lossi L, Ferrini F, Betelli C, Bardoni R. BDNF as a pain modulator. Prog Neurobiol. 2008 Jul;85(3):297-317. doi: 10.1016/j.pneurobio.2008.04.004. Epub 2008 Apr 26. PMID 18514997
- [Background] Obata K, Noguchi K. BDNF in sensory neurons and chronic pain. Neurosci Res. 2006 May;55(1):1-10. doi: 10.1016/j.neures.2006.01.005. Epub 2006 Mar 3. PMID 16516994
- [Background] Binder DK, Scharfman HE. Brain-derived neurotrophic factor. Growth Factors. 2004 Sep;22(3):123-31. doi: 10.1080/08977190410001723308. PMID 15518235
- [Background] Ritter AM, Lewin GR, Kremer NE, Mendell LM. Requirement for nerve growth factor in the development of myelinated nociceptors in vivo. Nature. 1991 Apr 11;350(6318):500-2. doi: 10.1038/350500a0. PMID 2014050
- [Background] Snider WD. Functions of the neurotrophins during nervous system development: what the knockouts are teaching us. Cell. 1994 Jun 3;77(5):627-38. doi: 10.1016/0092-8674(94)90048-5. No abstract available. PMID 8205613
- [Background] Woolf CJ, Safieh-Garabedian B, Ma QP, Crilly P, Winter J. Nerve growth factor contributes to the generation of inflammatory sensory hypersensitivity. Neuroscience. 1994 Sep;62(2):327-31. doi: 10.1016/0306-4522(94)90366-2. PMID 7530342
- [Background] Nicol GD, Vasko MR. Unraveling the story of NGF-mediated sensitization of nociceptive sensory neurons: ON or OFF the Trks? Mol Interv. 2007 Feb;7(1):26-41. doi: 10.1124/mi.7.1.6. PMID 17339604
- [Background] McKelvey L, Shorten GD, O'Keeffe GW. Nerve growth factor-mediated regulation of pain signalling and proposed new intervention strategies in clinical pain management. J Neurochem. 2013 Feb;124(3):276-89. doi: 10.1111/jnc.12093. PMID 23157347
- [Background] Miller RE, Malfait AM, Block JA. Current status of nerve growth factor antibodies for the treatment of osteoarthritis pain. Clin Exp Rheumatol. 2017 Sep-Oct;35 Suppl 107(5):85-87. Epub 2017 Sep 28. PMID 28967370

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pain Informed Movement
Started | 19 (19 is the number of participants enrolled in the study. 19 participants consented to participate and started the study.)
Completed | 14 (14 is the number of participants that stayed in the program and completed it.)
Not Completed | 5
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Arm/Group | Pain Informed Movement
Number analyzed (Participants) | 19
Age, Continuous [Mean (Full Range); unit: years] | 63.3 [48.0 to 84.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
BMI (kg/m^2) [Mean (Full Range); unit: kg/m^2] | 30.50 [20.32 to 42.04]

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Content
Description: A Likert scale out of 5 will assess how useful participants found the treatment. The minimum value is 1 and the maximum value is 5, with higher scores indicating a better outcome. The count of participants that reported the acceptability of content >4/5 is reported and considered for proceeding with the study without protocol amendment.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pain Informed Movement
Number analyzed (Participants) | 14
Participants | 13

2. Primary Outcome: Acceptability of Frequency
Description: A Likert scale out of 5 will assess how acceptable participants found the frequency of the treatment. The minimum value is 1 and the maximum value is 5, with higher scores indicating a better outcome. The count of participants that reported the acceptability of frequency >4/5 is reported and considered for proceeding with the study without protocol amendment.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pain Informed Movement
Number analyzed (Participants) | 14
Participants | 13

3. Primary Outcome: Acceptability of Duration
Description: A Likert scale out of 5 will assess how acceptable participants found the duration of the treatment. The minimum value is 1 and the maximum value is 5, with higher scores indicating a better outcome. The count of participants that reported the acceptability of duration >4/5 is reported and considered for proceeding with the study without protocol amendment.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pain Informed Movement
Number analyzed (Participants) | 14
Participants | 11

4. Primary Outcome: Burden of Questionnaires
Description: A numeric rating scale out of 10 will assess how burdensome participants found completing the questionnaires. On this scale,1 represents no burden at all and 10 represents very much a burden. Higher scores indicate a worse outcome. There is no minimum or maximum value. The count of participants that reported the burden <3/10 is reported and considered for proceeding with the study without protocol amendment
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pain Informed Movement
Number analyzed (Participants) | 14
Participants | 14

5. Primary Outcome: Burden of Physical Tests
Description: A numeric rating scale out of 10 will assess how burdensome participants found completing the physical tests. On this scale,1 represents no burden at all and 10 represents very much a burden. Higher scores indicate a worse outcome. The count of participants that reported the burden <3/10 is reported and considered for proceeding with the study without protocol amendment.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pain Informed Movement
Number analyzed (Participants) | 14
Participants | 14

6. Primary Outcome: Recruitment Rate
Description: Number of eligible participants who consent to participate in 1 month.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pain Informed Movement
Number analyzed (Participants) | 19
Participants | 19

7. Primary Outcome: Follow-Up Rate
Description: Percentage of participants who follow-up at 8 weeks.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pain Informed Movement
Number analyzed (Participants) | 19
Participants | 14

8. Primary Outcome: Self Reported Adverse Events
Description: Percentage of participants who did not experience any adverse events or only mild transient.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pain Informed Movement
Number analyzed (Participants) | 14
Participants | 14

9. Primary Outcome: Exercise Completion
Description: Percentage of participants who report exercising at least 3 times a week.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pain Informed Movement
Number analyzed (Participants) | 14
Participants | 13

10. Primary Outcome: Adherence
Description: Adherence to the program. This is the number of sessions that were attended by the participants. There are 2 sessions per week for 8 weeks, for a total of 16 sessions per participants. With 14 participants being in the study, the total number of sessions to be attended is 224. The number of sessions that were actually attended is being reported.
Time Frame: 8 weeks
Measure: Number; unit: sessions
Arm/Group | Pain Informed Movement
Number analyzed (Participants) | 14
sessions | 204

11. Primary Outcome: Recommending the Program
Description: Likelihood of recommending the program to others. On a scale of 1 to 5, participants rate how likely they would recommend the program to other people. On this scale, 1 is the minimum, and 5 is the maximum, with higher scores indicating a better outcome. Participants that indicate a score of 4 or 5 are counted as the number of participants that would likely recommend the program to others (the number being reported).
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pain Informed Movement
Number analyzed (Participants) | 14
Participants | 13

12. Primary Outcome: Using the Treatment Again
Description: Likelihood of using the treatment again. On a scale of 1 to 5, participants rate how likely they would use the treatment again. On this scale, 1 is the minimum, and 5 is the maximum, with higher scores indicating a better outcome. Participants that indicate a score of 4 or 5 are counted as the number of participants that would likely use it again (the number being reported).
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pain Informed Movement
Number analyzed (Participants) | 14
Participants | 13

13. Secondary Outcome: Change in Pain Modulation
Description: Pain modulation is assessed through conditioned pain modulation (CPM). First an ascending measure of pressure pain threshold (PPT) inducing a pain rating of 3/10 will be evaluated at the anterior shin on the unaffected knee. Next a conditioning stimulus in the form of forearm ischemia will be applied to induce a minimum verbal pain rating of 5/10 at the opposite volar forearm. Systolic pressure will be determined. The cuff will be inflated to 20mmhg above systolic pressure and the participant will be asked to squeeze a stress ball until a pain rating of 5/10 is reported. Once pain rating is recorded, PPT at the anterior shin will be repeated as the cuff remains inflated. An index will be created by calculating the percent efficiency of CPM (%CPM) as PPT2/PPT1, multiplied by 100; whereby %CPM ≤ 100 indicates inefficient pain modulation CPM. There is no minimum or maximum value. A change between two time points (baseline and 8 weeks) is reported.
Time Frame: Baseline, 8 weeks
Measure: Mean (Full Range); unit: Percentage of CPM
Arm/Group | Pain Informed Movement
Number analyzed (Participants) | 14
Percentage of CPM | 0.28 [-18.76 to 18.21]

14. Secondary Outcome: Change in Pain Intensity - Past 24 Hours
Description: Pain intensity will be measured using the numeric rating scale. Questions are rated on a an 11-point scale where patients select a rating between 0 and 10 with zero representing 'no pain' while 10 represents the 'worst imaginable pain. Higher scores mean a worse outcome. A change between two time points (baseline and 8 weeks) is reported.
Time Frame: Baseline, 8 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Pain Informed Movement
Number analyzed (Participants) | 14
score on a scale | -1.86 [-2.79 to -0.93]

15. Secondary Outcome: Change in Function
Description: Function will be measured using the Knee Injury and Osteoarthritis Outcome Score. The Knee Injury and Osteoarthritis Outcome Score has 42 items in 5 scored sub scales, of which two will be used: 1) pain, and 2) function in daily living (ADL). Scores range from 0-100 with zero representing extreme knee problems and 100 representing no knee problems. Higher scores mean a better outcome. A change between two time points (baseline and 8 weeks) is reported.
Time Frame: 8 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Pain Informed Movement
Number analyzed (Participants) | 14
score on a scale | 24.86 [14.46 to 36.27]

16. Secondary Outcome: Change in Brain-derived Neurotrophic Factor
Description: Brain-derived neurotrophic factor is a neurotrophin that appears to play a role in the central modulation of pain and pathophysiology of chronic pain. Blood will be drawn for analysis of brain-derived neurotrophic factor reported in ng/ml. There is no minimum or maximum values. A change between two time points (baseline and 8 weeks) is reported.
Time Frame: 8 weeks
Measure: Mean (95% Confidence Interval); unit: ng/ml
Arm/Group | Pain Informed Movement
Number analyzed (Participants) | 14
ng/ml | -2.36 [-7.77 to 3.04]

17. Secondary Outcome: Change in Pain Catastrophizing
Description: Pain catastrophizing scale will be measuring pain catastrophizing. It is a 13-item self reporting instrument. Each item on the scale is rated on a 5-point scale, ranging from 0 (not at all) to 4 (all the time). The total score on the PCS is the sum of the ratings for all 13 items, ranging from 0 to 52, with higher scores indicating higher pain catastrophizing (worse outcome). Subscales are combined to get the total score. Sub-scores for 3 dimensions will be used - rumination (range 0 to 12), magnification (range 0 to 12), and helplessness (range 0 to 28). A change between two time points (baseline and 8 weeks) is reported.
Time Frame: 8 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Pain Informed Movement
Number analyzed (Participants) | 14
score on a scale | -6.79 [-10.93 to -2.64]

18. Secondary Outcome: Change in Chronic Pain Self-efficacy
Description: Self-Efficacy for Managing Chronic Disease is a 6-item scale. The minimum value on each item is 1 and the maximum value on each item is 10. The score for the scale is the mean of the six items. The range for the total score is 1 to 10, with higher scores indicating higher self-efficacy and mean a better outcome. A change between two time points (baseline and 8 weeks) is reported.
Time Frame: 8 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Pain Informed Movement
Number analyzed (Participants) | 14
score on a scale | 1.54 [0.09 to 2.98]

19. Secondary Outcome: Change in Physical Performance Tests
Description: The 30 Second Sit to Stand Test will be used to test leg strength and endurance. The maximum number of chair stand repetitions completed during a 30 second interval will be noted along with use of any aids during testing. A change between two time points (baseline and 8 weeks) is reported.
Time Frame: 8 weeks
Measure: Mean (95% Confidence Interval); unit: Numbers of sit to stands
Arm/Group | Pain Informed Movement
Number analyzed (Participants) | 14
Numbers of sit to stands | 4.71 [3.09 to 6.34]

20. Secondary Outcome: Change in Anxiety and Depression
Description: Hospital Anxiety and Depression Scale consists of 7 questions to measure anxiety and 7 questions to measure depression. The minimum value on each item is 0 and the maximum value on each item is 3. The total score range is 0 to 21 for each subscale and higher scores represent increased severity in anxiety and depression symptoms (worse outcome). A total score can be created by combining the two subscales and the range would be from 0 to 42. A change between two time points (baseline and 8 weeks) is reported.
Time Frame: 8 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Pain Informed Movement
Number analyzed (Participants) | 14
score on a scale | 0.43 [-3.73 to 4.58]

21. Secondary Outcome: Change in Perspectives on Knee Replacement Surgery 1
Description: The question being asked is: Are your knee symptoms so severe that you wish to undergo knee replacement surgery? Answer options are yes, no, or unsure. There is no minimum, maximum, or total score. Count of participants that report Yes are reported.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pain Informed Movement
Number analyzed (Participants) | 14
Participants | 4

22. Secondary Outcome: Change in Perspectives on Knee Replacement Surgery 2
Description: The question being asked is: Do you think knee replacement surgery is eventually inevitable? Answer options are yes or no. There is no minimum, maximum, or total score. Count of participants that report Yes are reported.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pain Informed Movement
Number analyzed (Participants) | 14
Participants | 0

23. Secondary Outcome: Change in Perspectives on Knee Replacement Surgery 3
Description: The question being asked is: In your opinion, what factor(s) can lead to better outcomes after knee replacement surgery? Participants are given the following options to choose from: Good surgeon, healthy weight, good overall health, good social support, good mental health, less pain and disability before the surgery due to regular exercise, good hospital, not working (including house work), using pain killers after the surgery. Count of participants that do not choose 'less pain and disability before the surgery due to regular exercise' is reported.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pain Informed Movement
Number analyzed (Participants) | 14
Participants | 3

24. Secondary Outcome: Change in Pain
Description: Pain will also be measured using the Knee Injury and Osteoarthritis Outcome Score. The Knee Injury and Osteoarthritis Outcome Score has 42 items in 5 scored sub scales, of which two will be used: 1) pain, and 2) function in daily living (ADL). Scores range from 0-100 with zero representing extreme knee problems and 100 representing no knee problems (better outcome). A change between two time points (baseline and 8 weeks) is reported.
Time Frame: 8 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Pain Informed Movement
Number analyzed (Participants) | 14
score on a scale | 21.77 [11.24 to 32.30]

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Pain Informed Movement
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

LIMITATIONS AND CAVEATS:
Modification of inclusion criteria needed for future pilot RCT to enhance recruitment process.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-07): https://cdn.clinicaltrials.gov/large-docs/86/NCT04954586/Prot_SAP_000.pdf